CLINICAL TRIAL: NCT00259935
Title: A Study to Determine the Bioequivalence of an Oral Formulation of Topotecan Containing the Drug Substance Manufactured by New Process Relative to the Current Study Formulation of Topotecan in Patients With Advanced Solid Tumors (4C)
Brief Title: A Study To Determine If Two Different Versions Of Topotecan Have The Same Potency In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 104864/692
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer, Small Cell
Keywords: Any Solid Tumor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All treated subjects (Experimental): Subjects were randomized to receive 4 mg of a new formulation and current formulation of oral topotecan on Days 1 and 8 of Course 1.
  Interventions: Drug: topotecan

INTERVENTIONS:
Drug: topotecan — topotecan

SUMMARY:
The purpose of this study is to determine the bioequivalence of the new oral capsule formulation to the currently used oral capsule formulation of topotecan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced solid tumors.
* At least 4 weeks since last chemotherapy, radiotherapy, biologic therapy or surgery.
* Subjects must be free of post-treatment side effects.

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects with uncontrolled emesis, regardless of etiology, active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2004-10-04 (Actual); Primary Completion 2007-07-05 (Actual); Study Completion 2007-07-05 (Actual)

PRIMARY OUTCOMES:
Comparison of blood levels of topotecan following oral and IV dosing; blood samples will be drawn on Day 1 and Day 8 of Courses 1 and 2. | Days 1, 8

SECONDARY OUTCOMES:
Assessment of clinical laboratory tests, cardiac monitoring and disease progression. Comparison of blood levels of topotecan when taken orally with and without food; blood samples will be drawn on Day 1 | Up to 38 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (6):
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Morgantown, West Virginia
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht

REFERENCES:
- See also: Results for study 104864/692 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/104864/692?search=study&study_ids=104864%2F692#rs